CLINICAL TRIAL: NCT01654536
Title: A 6 Month Randomized, Open Label, Parallel Group, Safety Study Of Ciclesonide Nasal Aerosol (Zetonna®) And Ciclesonide Nasal Spray (Omnaris®) In Subjects 12 Years And Older With Perennial Allergic Rhinitis
Brief Title: A 6 Month Safety Study Of Ciclesonide Nasal Aerosol (Zetonna®) And Ciclesonide Nasal Spray (Omnaris®) In Subjects 12 Years And Older With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEP060-401
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Perennial Allergic Rhinitis
Keywords: PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ciclesonide nasal aerosol (Experimental): ciclesonide nasal aerosol 74 mcg
  Interventions: Drug: ciclesonide nasal aerosol
- ciclesonide nasal spray (Active Comparator): ciclesonide nasal spray 200 mcg
  Interventions: Drug: ciclesonide nasal spray

INTERVENTIONS:
Drug: ciclesonide nasal aerosol — ciclesonide nasal aerosol 74 mcg (given as 1 actuation per nostril of 37 mcg ciclesonide nasal aerosol)
  Other Names: Zetonna
  Arms: ciclesonide nasal aerosol
Drug: ciclesonide nasal spray — ciclesonide nasal spray 200 mcg (given as 2 actuations per nostril of 50 mcg ciclesonide nasal spray)
  Other Names: Omnaris
  Arms: ciclesonide nasal spray

SUMMARY:
This is a 6 month, multicenter, randomized, open label, parallel group, study to evaluate the nasal safety of ciclesonide nasal aerosol and ciclesonide aqueous nasal spray administered once daily to male and female subjects 12 years and older diagnosed with PAR.

DETAILED DESCRIPTION:
This is a 6 month, multicenter, randomized, open label, parallel group, safety study of ciclesonide nasal aerosol and ciclesonide aqueous nasal spray administered once daily to male and female subjects 12 years and older diagnosed with PAR. The objectives of this study are to evaluate the nasal and ocular safety of once daily dosing with ciclesonide nasal aerosol (Zetonna) 74 mcg and ciclesonide aqueous nasal spray (Omnaris) 200 mcg in subjects 12 years and older with PAR.

ELIGIBILITY:
Inclusion Criteria:

* Subject or Subject's parent/guardian gives written informed consent and assent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Male or female 12 years and older, as of the Screening visit.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, medical history.
* A history of PAR to a relevant perennial allergen (eg, house dust mites, cockroach, molds, animal dander) for a minimum of one year immediately preceding the study Screening visit. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past 12 months, and require treatment throughout the entire study period.
* Subject, if female ≤ 65 years of age, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

  * An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation.
  * Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  * Abstinence.
* Subject must possess an educational level and degree of understanding of English that enables them to communicate suitably with the PI and study coordinator.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Current physical findings of nasal polyps, septal perforation, or nasal ulceration. (Subjects showing significant progression of nasal pathology between screening and randomization would be excluded at the discretion of the investigator.]
* Planned insertion of nasal septal jewelry during the study period.
* Surgery (including biopsy) and atrophic rhinitis or rhinitis medicamentosa are not permitted within the last 30 days prior to the Screening visit.
* Participation in any investigational drug trial within the 30 days preceding the Screening visit or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening visit.
* History of alcohol or drug abuse within 2 years preceding the Screening visit.
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Active asthma requiring treatment with inhaled or systemic corticosteroids.
* Use of chronic treatment with agents known to promote the development of cataracts (potassium-sparing diuretics and allopurinol).
* Non vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit.
* Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Use of nasal corticosteroids within 14 days, or ocular, oral or parenteral within 6 months prior to randomization.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial:

  1. impaired hepatic function including alcohol related liver disease or cirrhosis
  2. diabetes mellitus
  3. malignancy (excluding basal cell carcinoma)
* Any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written Ocular Exclusion Criteria
* History of bacterial or viral infection of the eyes within 14 days of the Screening visit or current or history of ocular herpes simplex.
* Any use within 6 months prior to the randomization or planned use during the trial of a topical ocular corticosteroid, or intraocular or periocular injection of corticosteroids.
* Progressive retinal (including, but not limited to acute macular degeneration or unstable diabetic retinopathy) or optic nerve disease in either eye.
* Ocular injury/surgery in the last 6 months (including LASIK eye surgery, as well as any glaucoma intraocular surgery, including laser trabeculoplasty [ALT or SLT]).
* Any evidence of glaucomatous optic disc changes or a vertical cup:disc ratio > 0.8.
* Current or history of any glaucoma related diagnosis, including ocular hypertension, open-angle or closed-angle, as well as secondary or congenital glaucoma.
* Occludable angles by slit lamp examination (eg, peripheral anterior chamber less than or equal to one quarter of the peripheral corneal thickness), which may be confirmed by gonioscopy at the investigator's discretion..
* Current PSC cataract or previous history of cataract surgery.
* Current or history of congenital cataract or active or prior uveitis.
* Historical or current intraocular pressure of 22 mm Hg or higher in either eye.
* Inability to complete ocular examination, including: Inability to measure intraocular pressure, Pupillary diameter < 6 mm upon dilation , Significant media opacity in either eye that would exclude adequate posterior segment examination, Clinically significant corneal dystrophy, epithelial, or endothelial disease that would preclude visualization or intraocular pressure measurement, Corneal irregularities or scarring that in the investigator's judgment would impeded an accurate measurement of intraocular pressure or visualization of intraocular anatomy, Unwillingness to remove contact lenses for ocular examination, Subjects with LOCS III grade NO > 4.0, NC > 4.0 and C > 4.0 in either eye
* Best-corrected visual acuity in either eye of 20/200 or worse at the screening ocular examination.
* Planned or anticipated ocular surgery during the next 6 months.
* Any condition that, in the judgment of the ophthalmologist, would preclude the subject from completing the protocol with capture of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (31):
- United States (31):
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - CHOC PSF AMC - Division of Allergy, Asthma and Immunology, Orange, California
  - Allergy Associates Medical Group Inc., San Diego, California
  - Bensch Research Associates, Stockton, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - DataQuest Medical Research LLC, Lawerenceville, Georgia
  - Asthma & Allergy Consultants, PC, Lilburn, Georgia
  - Gordon D Raphael, MD, Bethesda, Maryland
  - Medical Education and Research Management Services of New England, Gardner, Massachusetts
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Clinical Research Institute Inc., Minneappolis, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Clinical Research Group of Montanta, Bozeman, Montana
  - Ocean Allergy & Respiratory Research Center, Brick, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Allergy and Asthma Center of NC, PA, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy Assocaites Research Center, Portland, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - National Allergy, Asthma & Uticaria Centers of Charleston, P.A., Charleston, South Carolina
  - Isis Clinical Research, LLC, Austin, Texas
  - Sirius Clinical Research LLC, Austin, Texas
  - Pharmaceutical Research and Consulting Inc., Dallas, Texas
  - Kerrville Research Associates, PA, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - ASTHMA Inc. Clinical Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciclesonide Nasal Aerosol: Zetonna (ciclesonide) nasal aerosol 74 mcg
  ciclesonide nasal aerosol: ciclesonide nasal aerosol 74 mcg (given as 1 actuation per nostril of 37 mcg ciclesonide nasal aerosol)
- Ciclesonide Nasal Spray: Omnaris (ciclesonide) nasal spray 200 mcg
  ciclesonide nasal spray: ciclesonide nasal spray 200 mcg (given as 2 actuations per nostril of 50 mcg ciclesonide nasal spray)
Period: Overall Study
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Started | 368 | 369
Completed | 324 | 331
Not Completed | 44 | 38
Not completed — Lost to Follow-up | 5 | 5
Not completed — Physician Decision | 12 | 8
Not completed — Withdrawal by Subject | 27 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray | Total
Number analyzed (Participants) | 368 | 369 | 737
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 43 | 83
  Between 18 and 65 years | 322 | 321 | 643
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.09) | 37.7 (14.03) | 37.8 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 235 | 482
  Male | 121 | 134 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 53 | 105
  Not Hispanic or Latino | 315 | 314 | 629
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 69 | 58 | 127
  White | 272 | 289 | 561
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 368 | 369 | 737

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Experiencing Nasal Mucosal Disorders, Septum Disorders, or Nasal Septum Perforations as Treatment Emergent Adverse Events (AEs; TEAE)
Time Frame: 0-6 months
Population: Safety Population: The safety population consisted of all randomly assigned subjects who received at least 1 dose of study medication. The safety population was expected to be the same as the ITT population. However, if there were any subjects who were mis randomized, the actual treatment taken would have been used for the analyses.
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants
  Any Nasal Mucosal Disorder, Septum Disorder, or Na | 3 | 4
  Nasal Mucosal Disorder | 2 | 0
  Nasal Septum Disorder | 0 | 0
  Nasal Septum Ulceration | 1 | 4
  Nasal Septum Perforation | 0 | 0

2. Secondary Outcome: The Number of Subjects Experiencing Treatment Emergent Nasal AEs.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants
  Overall | 53 | 44
  General Disorders and Administration Site Conditio | 5 | 0
  Application site pain | 5 | 0
  Infections and Infestations | 11 | 8
  Acute sinusitis | 1 | 1
  Sinusitis | 10 | 7
  Injury, Poisoning and Procedural Complications | 2 | 2
  Facial bones fracture | 0 | 1
  Mucosal excoriation | 0 | 1
  Scratch | 2 | 0
  Nervous System Disorders | 0 | 1
  Sinus headache | 0 | 1
  Respiratory, Thoracic and Mediastinal Disorders | 41 | 34
  Epistaxis | 22 | 26
  Nasal congestion | 4 | 2
  Nasal discomfort | 6 | 4
  Nasal dryness | 1 | 1
  Nasal mucosal discolouration | 0 | 1
  Nasal mucosal disorder | 2 | 0
  Nasal septum ulceration | 1 | 4
  Paranasal sinus hypersecretion | 2 | 1
  Respiratory tract congestion | 1 | 0
  Rhinalgia | 2 | 0
  Rhinorrhoea | 2 | 0
  Sinus congestion | 3 | 1
  Sneezing | 6 | 0
  Skin and Subcutaneous Tissue Disorders | 0 | 1
  Scab | 0 | 1

3. Secondary Outcome: The Percentage of Subjects Experiencing Treatment Emergent Nasal AEs.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants
  Overall | 14.4 | 11.9
  General Disorders and Administration Site Conditio | 1.4 | 0
  Application site pain | 1.4 | 0
  Infections and Infestations | 3.0 | 2.2
  Acute sinusitis | 0.3 | 0.3
  Sinusitis | 2.7 | 1.9
  Injury, Poisoning and Procedural Complications | 0.5 | 0.5
  Facial bones fracture | 0 | 0.3
  Mucosal excoriation | 0 | 0.3
  Scratch | 0.5 | 0
  Nervous System Disorders | 0 | 0.3
  Sinus headache | 0 | 0.3
  Respiratory, Thoracic and Mediastinal Disorders | 11.2 | 9.2
  Epistaxis | 6.0 | 7.0
  Nasal congestion | 1.1 | 0.5
  Nasal discomfort | 1.6 | 1.1
  Nasal dryness | 0.3 | 0.3
  Nasal mucosal discolouration | 0 | 0.3
  Nasal mucosal disorder | 0.5 | 0
  Nasal septum ulceration | 0.3 | 1.1
  Paranasal sinus hypersecretion | 0.5 | 0.3
  Respiratory tract congestion | 0.3 | 0
  Rhinalgia | 0.5 | 0
  Rhinorrhoea | 0.5 | 0
  Sinus congestion | 0.8 | 0.3
  Sneezing | 1.6 | 0
  Skin and Subcutaneous Tissue Disorders | 0 | 0.3
  Scab | 0 | 0.3

4. Secondary Outcome: The Number of Subjects Experiencing Treatment Emergent AEs.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants
  Overall | 121 | 114
  General Disorders and Administration Site Conditio | 7 | 3
  Application site pain | 5 | 0
  Infections and Infestations | 55 | 46
  Bronchitis | 5 | 3
  Gastroenteritis viral | 6 | 0
  Influenza | 7 | 3
  Nasopharyngitis | 12 | 11
  Sinusitis | 10 | 7
  Upper respiratory tract infection | 12 | 8
  Viral upper respiratory tract infection | 5 | 5
  Injury, Poisoning and Procedural Complications | 11 | 13
  Muscle strain | 0 | 4
  Nervous System Disorders | 9 | 14
  Headache | 4 | 9
  Respiratory, Thoracic and Mediastinal Disorders | 49 | 37
  Asthma | 4 | 1
  Cough | 4 | 2
  Epistaxis | 22 | 26
  Nasal congestion | 4 | 2
  Nasal discomfort | 6 | 4
  Nasal septum ulceration | 1 | 4
  Sneezing | 6 | 0

5. Secondary Outcome: The Percentage of Subjects Experiencing Treatment Emergent AEs.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants
  Overall | 33.0 | 30.8
  General Disorders and Administration Site Conditio | 1.9 | 0.8
  Application site pain | 1.4 | 0
  Infections and Infestations | 15.0 | 12.4
  Bronchitis | 1.4 | 0.8
  Gastroenteritis viral | 1.6 | 0
  Influenza | 1.9 | 0.8
  Nasopharyngitis | 3.3 | 3.0
  Sinusitis | 2.7 | 1.9
  Upper respiratory tract infection | 3.3 | 2.2
  Viral upper respiratory tract infection | 1.4 | 1.4
  Injury, Poisoning and Procedural Complications | 3.0 | 3.5
  Muscle strain | 0 | 1.1
  Nervous System Disorders | 2.5 | 3.8
  Headache | 1.1 | 2.4
  Respiratory, Thoracic and Mediastinal Disorders | 13.4 | 10.0
  Asthma | 1.1 | 0.3
  Cough | 1.1 | 0.5
  Epistaxis | 6.0 | 7.0
  Nasal congestion | 1.1 | 0.5
  Nasal discomfort | 1.6 | 1.1
  Nasal septum ulceration | 0.3 | 1.1
  Sneezing | 1.6 | 0

6. Secondary Outcome: The Number of Subjects Experiencing Treatment Emergent Serious Adverse Events (SAEs).
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Ciclesonide Nasal Aerosol: Zetona (ciclesonide) nasal aerosol 74 mcg
  ciclesonide nasal aerosol: ciclesonide nasal aerosol 74 mcg (given as 1 actuation per nostril of 37 mcg ciclesonide nasal aerosol)
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants
  Overall | 4 | 5
  Cardiac Disorders | 0 | 1
  Angina pectoris | 0 | 1
  Coronary artery disease | 0 | 1
  Hepatobiliary Disorders | 0 | 1
  Bile duct stenosis | 0 | 1
  Infections and Infestations | 0 | 1
  Appendicitis | 0 | 1
  Injury, Poisoning and Procedural Complications | 1 | 1
  Facial bones fracture | 0 | 1
  Limb injury | 1 | 0
  Investigations | 0 | 1
  Blood pressure increased | 0 | 1
  Nervous System Disorders | 2 | 0
  Lacunar infarction | 1 | 0
  Migraine | 1 | 0
  Reproductive System and Breast Disorders | 0 | 1
  Postmenopausal haemorrhage | 0 | 1
  Respiratory, Thoracic and Mediastinal Disorders | 1 | 0
  Pulmonary embolism | 1 | 0

7. Primary Outcome: The Percentage of Subjects Experiencing Nasal Mucosal Disorders, Septum Disorders, or Nasal Septum Perforations as Treatment Emergent Adverse Events (AEs; TEAE)
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants
  Any Nasal Mucosal Disorder, Septum Disorder, or Na | 0.8 | 1.1
  Nasal Mucosal Disorder | 0.5 | 0
  Nasal Septum Disorder | 0 | 0
  Nasal Septum Ulceration | 0.3 | 1.1
  Nasal Septum Perforation | 0 | 0

8. Secondary Outcome: The Percentage of Subjects Experiencing Treatment Emergent Serious Adverse Events (SAEs).
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants
  Overall | 1.1 | 1.4
  Cardiac Disorders | 0 | 0.3
  Angina pectoris | 0 | 0.3
  Coronary artery disease | 0 | 0.3
  Hepatobiliary Disorders | 0 | 0.3
  Bile duct stenosis | 0 | 0.3
  Infections and Infestations | 0 | 0.3
  Appendicitis | 0 | 0.3
  Injury, Poisoning and Procedural Complications | 0.3 | 0.3
  Facial bones fracture | 0 | 0.3
  Limb injury | 0.3 | 0
  Investigations | 0 | 0.3
  Blood pressure increased | 0 | 0.3
  Nervous System Disorders | 0.5 | 0
  Lacunar infarction | 0.3 | 0
  Migraine | 0.3 | 0
  Reproductive System and Breast Disorders | 0 | 0.3
  Postmenopausal haemorrhage | 0 | 0.4
  Respiratory, Thoracic and Mediastinal Disorders | 0.3 | 0
  Pulmonary embolism | 0.3 | 0

9. Secondary Outcome: The Number of Subjects Experiencing Treatment Emergent AEs Causing Study Medication Discontinuation.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants
  Overall | 13 | 12
  Cardiac Disorders | 0 | 1
  Angina pectoris | 0 | 1
  Coronary artery disease | 0 | 1
  Ear and Labyrinth Disorders | 1 | 1
  Ear pain | 1 | 0
  Tinnitus | 0 | 1
  Eye Disorders | 1 | 0
  Vision blurred | 1 | 0
  Infections and Infestations | 3 | 1
  Bronchitis | 1 | 0
  Pelvic inflammatory disease | 1 | 0
  Upper respiratory tract infection | 1 | 1
  Injury, Poisoning and Procedural Complications | 0 | 2
  Facial bones fracture | 0 | 1
  Mucosal excoriation | 0 | 1
  Investigations | 1 | 1
  Blood pressure increased | 0 | 1
  Intraocular pressure increased | 1 | 0
  Nervous System Disorders | 3 | 2
  Dizziness | 0 | 1
  Headache | 2 | 1
  Lacunar infarction | 1 | 0
  Nerve compression | 1 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 7 | 5
  Asthma | 2 | 1
  Epistaxis | 1 | 3
  Nasal congestion | 0 | 1
  Nasal discomfort | 2 | 1
  Pulmonary embolism | 1 | 0
  Sneezing | 1 | 0
  Skin and Subcutaneous Tissue Disorders | 0 | 1
  Urticaria | 0 | 1
  Vascular Disorders | 0 | 1
  Haematoma | 0 | 1

10. Secondary Outcome: The Percentage of Subjects Experiencing Treatment Emergent AEs Causing Study Medication Discontinuation.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants
  Overall | 3.5 | 3.2
  Cardiac Disorders | 0 | 0.3
  Angina pectoris | 0 | 0.3
  Coronary artery disease | 0 | 0.3
  Ear and Labyrinth Disorders | 0.3 | 0.3
  Ear pain | 0.3 | 0
  Tinnitus | 0 | 0.3
  Eye Disorders | 0.3 | 0
  Vision blurred | 0.3 | 0
  Infections and Infestations | 0.8 | 0.3
  Bronchitis | 0.3 | 0
  Pelvic inflammatory disease | 0.3 | 0
  Upper respiratory tract infection | 0.3 | 0.3
  Injury, Poisoning and Procedural Complications | 0 | 0.5
  Facial bones fracture | 0 | 0.3
  Mucosal excoriation | 0 | 0.3
  Investigations | 0.3 | 0.3
  Blood pressure increased | 0 | 0.3
  Intraocular pressure increased | 0.3 | 0
  Nervous System Disorders | 0.8 | 0.5
  Dizziness | 0 | 0.3
  Headache | 0.5 | 0.3
  Lacunar infarction | 0.3 | 0
  Nerve compression | 0.3 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 1.9 | 1.4
  Asthma | 0.5 | 0.3
  Epistaxis | 0.3 | 0.8
  Nasal congestion | 0 | 0.3
  Nasal discomfort | 0.5 | 0.3
  Pulmonary embolism | 0.3 | 0
  Sneezing | 0.3 | 0
  Skin and Subcutaneous Tissue Disorders | 0 | 0.3
  Urticaria | 0 | 0.3
  Vascular Disorders | 0 | 0.3
  Haematoma | 0 | 0.3

11. Secondary Outcome: Number of Subjects With Development of or Worsening in Lens Opacities.
Time Frame: 0-6 months
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants | 51 | 53

12. Secondary Outcome: Percentage of Subjects With Development of or Worsening in Lens Opacities.
Time Frame: 0-6 months
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants | 13.9 | 14.3

13. Secondary Outcome: Number of Subjects With Increase ≥ 7 mm Hg From Baseline in Intraocular Pressure, or a Change to > 21 mm Hg, in Either Eye
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants | 9 | 6

14. Secondary Outcome: Percentage of Subjects With Increase ≥ 7 mm Hg From Baseline in Intraocular Pressure, or a Change to > 21 mm Hg, in Either Eye
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of partcipants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of partcipants | 2.5 | 1.6

15. Secondary Outcome: Number of Subjects With Change From Baseline in Best Corrected Visual Acuity.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
participants | 1 | 2

16. Secondary Outcome: Percentage of Subjects With Change From Baseline in Best Corrected Visual Acuity.
Time Frame: 0-6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Number analyzed (Participants) | 367 | 370
percentage of participants | 0.3 | 0.5

ADVERSE EVENTS:
Time Frame: 0-6 months
Description: Safety Population: The safety population consisted of all randomly assigned subjects who received at least 1 dose of study medication. The safety population was expected to be the same as the ITT population. However, if there were any subjects who were mis randomized, the actual treatment taken would have been used for the analyses.
Arm/Group | Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray
Serious Adverse Events (participants affected / at risk) | 4/367 | 5/370
Other Adverse Events (participants affected / at risk) | 22/367 | 26/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide Nasal Aerosol (N=367) | Ciclesonide Nasal Spray (N=370)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure (Investigations) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage* (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide Nasal Aerosol (N=367) | Ciclesonide Nasal Spray (N=370)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.